CLINICAL TRIAL: NCT02030899
Title: The Comparison Between the Stand-alone Cage and the Autologous Iliac Bone Graft/Anterior Plating in the Single-level Surgical Treatment of the Cervical Spine
Acronym: CAP_2014
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chun Kee Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP_2014
Record Dates: First submitted 2014-01-02; First posted 2014-01-09 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cervical Vertebrae; Single; Degenerative Disease
Keywords: Cervical vertebrae; single; degenerative disease; Fusion; Sagittal angle

STUDY DESIGN:
Intervention Model Description: ACDF with plate and autologous bone
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cage (Active Comparator): Cage filled with autologous bone
  Interventions: Procedure: Cage fusion
- Plate (Other): Plate augmentation after iliac bone graft
  Interventions: Procedure: Plate fusion

INTERVENTIONS:
Procedure: Cage fusion — Randomized selection of surgery type
  Other Names: Use of stand-alone Cage filled with autologous bone
  Arms: Cage
Procedure: Plate fusion — Randomized selection of surgery type
  Other Names: Use of Plate augmentation after autologous iliac bone graft
  Arms: Plate

SUMMARY:
The use of plate in addition to autologous bone is better then stand alone cage fusion regarding fusion rate and segmental lordosis.

DETAILED DESCRIPTION:
cage: MC+® cage plate: atlantis® plate

ELIGIBILITY:
Inclusion Criteria:

* Single level degenerative cervical spine disease
* aged 30 - 70
* no improvement of symptom for 8 weeks of non-surgical treatment.
* degeneration in other levels without stenosis, accepted

Exclusion Criteria:

* osteoporosis
* disease with poor bone quality
* Cancer
* Previous cervical spine surgery
* Multiple levels disease
* Ossification of posterior longitudinal ligament
* Kyphosis at the index level
* Developmental stenosis (diameter of C7 spinal canal < 10mm)

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Fusion rate | 2 years
  The rate of interbody fusion at 2 years

SECONDARY OUTCOMES:
Segmental angle | 2 years
  the segmental angle at the fused level
cervical lordosis | 2 years
  The cervical lordosis at 2 years
pain change | 2 years
  Visual analogue pain score
functional status change. | 2 years
  Neck disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea